CLINICAL TRIAL: NCT02897375
Title: A Phase 1 Study of Palbociclib in Combination With Cisplatin or Carboplatin in Advanced Solid Malignancies
Brief Title: Palbociclib With Cisplatin or Carboplatin in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Olatunji Alese, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00089583; NCI-2016-01037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3263-16 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2016-08-30; First posted 2016-09-13 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Solid Neoplasm; Stage III Pancreatic Cancer; Stage IIIA Breast Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Breast Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage IV Non-Small Cell Lung Cancer; Stage IVA Pancreatic Cancer; Stage IVB Pancreatic Cancer; Sarcoma; Colorectal Cancer; Head and Neck Cancer; Cancer of Unknown Primary; Bladder Cancer; Ovarian Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Sarcoma; Colorectal Neoplasms; Head and Neck Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Cisplatin; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (palbociclib, cisplatin) (Experimental): Patients receive cisplatin IV over 30-60 minutes on day 1 and palbociclib PO QD on days 2-22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Palbociclib
- Arm B (palbociclib, carboplatin) (Experimental): Patients receive carboplatin IV over 30-60 minutes on day 1 and palbociclib PO QD on days 2-22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Palbociclib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Paraplatin
  Arms: Arm B (palbociclib, carboplatin)
Drug: Cisplatin — Given IV
  Other Names: CDDP; Cis-diamminedichloridoplatinum; Cisplatinum; Cismaplat; Neoplatin
  Arms: Arm A (palbociclib, cisplatin)
Drug: Palbociclib — Given PO
  Other Names: Ibrance; PD-0332991

SUMMARY:
This phase I trial studies the side effects and best dose of palbociclib with cisplatin or carboplatin in treating patients with solid tumors that have spread to other places and usually cannot be cured or controlled with treatment. Palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving palbociclib with cisplatin or carboplatin may help stop tumor growth in patients with advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and tolerability of palbociclib when administered along with cisplatin or carboplatin.

II. Establish the recommended phase 2 dose (RP2D) of the tested combinations.

SECONDARY OBJECTIVES:

I. Characterize the pharmacokinetic (PK) profiles of cisplatin, carboplatin.

II. Obtain preliminary evidence of anti-tumor efficacy of the tested combination regimens.

III. Conduct PK/pharmacodynamics (PD) correlative analyses using palbociclib trough concentration and cyclin-dependent kinase 4 (CDK4) inhibition read-outs in tumor and surrogate samples collected on course 1 day 22 (C1D22).

IV. Assess potential association between tissue-based biomarkers and efficacy.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 arms.

ARM A: Patients receive cisplatin intravenously (IV) over 30-60 minutes on day 1 and palbociclib orally (PO) once daily (QD) on days 2-22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive carboplatin IV over 30-60 minutes on day 1 and palbociclib PO QD on days 2-22. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed solid organ malignancy
* Patients enrolled in the expansion cohort must have histologically or cytologically confirmed squamous non-small cell lung cancer (NSCLC), breast or pancreaticobiliary tract cancer
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) with conventional techniques or as ≥ 10 mm (≥ 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Leukocytes ≥ 3,000/mL
* Absolute neutrophil count ≥ 1,500/mL
* Platelets ≥ 100,000/mL
* Hemoglobin ≥ 10 g/dL
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (except for patients with Gilbert disease)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 × institutional upper limit of normal (up to 5 X upper limit of normal [ULN] for patients with liver metastasis)
* Creatinine within normal institutional limits OR creatinine clearance ≥ 60 mL/min/1.73 m² for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 6 months after completion of study drug administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had cytotoxic anticancer chemotherapy or immune checkpoint inhibitor within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or palliative radiation within 2 weeks (stereotactic radiation therapy [SRS] for brain metastasis within 48 hours) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients receiving cytotoxic agent as immunomodulatory therapy for a non neoplastic indication (e.g. methotrexate for rheumatoid arthritis) and who are unable to discontinue such agents within 2 weeks prior to starting treatment
* Oral targeted therapy within five days or five half-lives, whichever is longer, prior to initiating protocol therapy treatment
* Patients who are receiving any other investigational agents
* Use of strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors and inducers
* Patients with symptomatic uncontrolled brain metastases are excluded; (patients with stable treated or asymptomatic untreated brain metastasis not requiring glucocorticoids are allowed)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib, carboplatin or cisplatin
* Concurrent administration of strong inducers and inhibitors of CYP3A enzyme or CYP3A substrates with narrow therapeutic window
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring intravenous antibiotics at the time of treatment initiation
  * Symptomatic congestive heart failure (requiring hospital stay within the last 6 months)
  * Myocardial infarction within the last 6 months
  * Unstable angina pectoris, cardiac arrhythmia
  * Psychiatric illness
* Social situations or circumstances that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with palbociclib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Study completion, an average of 2 years
Incidence of dose limiting toxicities defined as grade 3 or higher toxicity | Up to 4 weeks
Recommended phase 2 dose (RP2D) as the highest doses of palbociclib and cisplatin or palbociclib and carboplatin | Study completion, an average of 2 years

SECONDARY OUTCOMES:
Overall response rate (complete response + partial response) assessed by Response Evaluation Criteria in Solid Tumors 1.1 criteria | Up to 3 years
  Will be summarized and presented along with 95% exact confidence intervals.
Pharmacokinetic (PK) characteristics of carboplatin including maximum concentration (Cmax) | Up to 4 weeks
  Within-subject and between-cohort comparisons of Cmax will be performed using Wilcoxon (non-parametric) test.
Pharmacokinetic (PK) characteristics of cisplatin including maximum concentration (Cmax) | Up to 4 weeks
  Within-subject and between-cohort comparisons of Cmax will be performed using Wilcoxon (non-parametric) test.

CONTACTS AND LOCATIONS:
Overall Officials: Olatunji B Alese, MD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alese OB, Harvey RD, Wu C, Hitron E, Collins H, Scott S, Steuer C, Bilen MA, Carthon BC, Switchenko JM, Ramalingam SS, Owonikoko TK. Phase I study of palbociclib with cisplatin or carboplatin in the management of patients with advanced pancreatic cancer. Oncologist. 2025 Oct 1;30(10):oyaf284. doi: 10.1093/oncolo/oyaf284. PMID 40973049

DOCUMENTS (1):
  • Informed Consent Form (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT02897375/ICF_000.pdf